CLINICAL TRIAL: NCT00209690
Title: Phase I/II Study of Docetaxel, Cisplatin and 5-fluorouracil(TPF) as 1st-line Chemotherapy in Patients With Metastatic Esophageal Cancer.
Brief Title: Phase I/II Study of TPF as First-line Chemotherapy in Patients With Metastatic Esophageal Cancer.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hokkaido Gastrointestinal Cancer Study Group (Other)
Collaborators: Hokkaido University Hospital (Other)
Responsible Party: Yoshito Komatsu / A vice-director,, Hokkaido Gastrointestina Cancer Study Group
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGCSG0305-1; TPF
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2010-05-26 (Estimated); Status verified 2010-05

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Docetaxel; Fluorouracil; Cisplatin; DCM-Dex-CDDP

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Taxotere; Drug: 5-FU; Drug: Briplatin

INTERVENTIONS:
Drug: Taxotere — X mg/m2, IV (in the vein) on day 1 of each 28 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: Docetaxel
Drug: 5-FU — 800 mg/m2, CIV (conti.in the vein) on day 1~4 of each 28 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: 5-Fluorouracil
Drug: Briplatin — 15 mg/m2, IV (in the vein) on day 1~4 of each 28 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: Cisplatin,CDDP

SUMMARY:
A phase I/II study is conducted to determine the maximum-tolerated dose (MTD), dose-limiting toxicity (DLT), and efficacy of a combination chemotherapy using docetaxel, cisplatin and 5-fluorouracil (TPF) in untreated patients with metastatic esophageal cancer. The usefulness of the this regimen is evaluated by response rate, median survival time, and progression free survival.

DETAILED DESCRIPTION:
Patients with untreated measurable metastatic esophageal cancer were included in this trial. Patients received this combination chemotherapy repeated every 28 days until progression disease. Starting dose (dose level 1) were docetaxel 50 mg/m2 on day 1, fixed dose intravenously cisplatin (15 mg/m2/day) and continuous infusion 5-FU (800 mg/m2/day) on day 1-4. DLT was defined as follows (according to NCI-CTC version 2.0); Grade 4 neutropenia lasting for more than 4days, Grade 4 anemia and thrombocytopenia, Grade 3 neutropenia accompanied fever (>38℃) , and Grade 3 non-hematological toxicity (except for nausea, appetite loss , general fatigue). Maximal Tolerated Dose (MTD) is determined when the incidence of critical toxicity exceeds 50% at a certain dose level. Response rate will be calculated according to RECIST criteria.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic or recurrent esophageal tumors with no previous treatment for advanced disease.(Except for small cell carcinoma)
* At least one measurable lesion according to the RECIST criteria. Minimum indicator lesion size: > 10 mm measured by spiral CT or >20mm measured by conventional techniques(Except for Phase I setting).
* Patients aged between 20 and 75 years, inclusive, at the time of acquisition of informed consent
* Patients with performance status(ECOG) 0 to 2
* Abnormal hematologic values (WBC ≥ 3.0 x 109/L, Hemoglobin ≥ 9.5g/dl, platelet count ≥ 100 x 109/L)
* Creatinine clearance ≥ 60 ml/min, Serum cleatinine ≤ 1.5mg/dl
* Serum bilirubin ≤ 1.5mg/dl. ALT, AST ≤ 2.5 x upper normal limit (or ≤ 3 x upper normal limit in the case of liver metastases)
* Patients who have not received cancer therapy (radiotherapy, chemotherapy or immunotherapy)
* Life expectancy ≥ 3 months
* Patients who have given written informed consent to participate in this study

Exclusion Criteria:

* Patients with active multiple cancers; or even if the multiple cancers are metachronous, have a disease-free period of less than 5 years (but excluding cancer in situ and skin cancer) (Except for Phase I setting)
* Serious, uncontrolled, concurrent infection(s) or illness(es)
* Patients with no serious concurrent complications (such as heart disease, Intestinal pneumonia)
* Patients with brain metastasis
* Patients receiving continuous administration of steroids
* Patients who have experienced serious drug allergy in the past
* Patients with retention of body fluid(pleural effusion, ascites, pericardial effusion) necessitating treatment
* Patients who are pregnant and lactating or hope to become pregnant during the study period
* Patients with prior Taxan treatment (Paclitaxel, Docetaxel)
* Patients with edema ≥ grade 2
* Others, patients judged by the investigator or subinvestigator to be inappropriate as subject

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2003-10; Primary Completion 2009-12 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Determine the DLT(Dose Limiting Toxicity) and MTD(Maximum Tolerated Dose) in Phase I setting. Determine the clinical response rate with Recommended dose in Phase II setting. | one year

SECONDARY OUTCOMES:
Determine the MST(Median Survival Time) and PFS(Progression Free Survival) in Phase II setting. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Masahiro Asaka, MD, PhD, Study Chair — Hokkaido Gastrointestinal Cancer Study Group
Locations (1):
- ・ Hokkaido University Hospital (Hokkaido University Graduate School of Medicine / School of Medicine), Sapporo, Hokkaido, Japan